PROTOCOL TITLE: Wood stove interventions and child respiratory infections in rural communities

ClinicalTrials.gov Number: NCT02240134

PRINCIPAL INVESTIGATOR(S): Curtis W. Noonan and Tony J. Ward, School of Public and Community Health Sciences, University of Montana, 406-243-4957, <a href="mailto:curtis.noonan@umontana.edu">curtis.noonan@umontana.edu</a>

RESEARCH LOCATION(S): University of Montana, Missoula, MT; University of New Mexico, Albuquerque, NM; University of Alaska, Fairbanks, AK

DOCUMENT DATE: November 11, 2015
PROTOCOL AND REVISION HISTORY:

| Version | Summary of Change |
|---|---|
| Approval | |
| Date, | |
| mm/dd/yyyy | |
| 12/23/2013 | Original protocol |
| 08/26/2014 | Amendment for approval of recruitment flyers and media |
| 09/22/2014 | The following changes were made in the parental permission form |
| | 1. We will collect data about your home and child during two, six-month |
| | winter periods. For the data about your home, we will conduct up to two visits in the first winter. |
| | 2. At each of these visits we will place devices in your home for up to 6 days |
| | to measure temperature and dust. |
| 10/27/2014 | Data collection protocols and forms |
| 12/23/2014 | Addition of wipe sample collection to assess nicotine in homes. |
| | Parental permission form revised to include: "Once per winter, we will collect |
| | a nicotine wipe sample from a surface in the home that is very rarely cleaned |
| | (e.g., top of a door jam)." |
| 05/21/2015 | Amendment for approval of recruitment materials |
| 06/22/2015 | Amendment for approval of social media and radio recruitment messages |
| 09/14/2015 | Amendment to add two question added to Child Symptom Questionnaire: |
| | Did anyone in the home miss work because of your child's illness? No Yes |
| | If yes, for how many days: |
| 10/02/2015 | Amendment to add two questions to Home Characteristics Questionnaire: |
| | Does anyone in the household smoke? No Yes |
| | If yes, do they smoke inside the home? No Yes |
| 11/11/2015 | Amendment to add End of Winter Home Questionnaires and Knowledge, Attitudes, Behaviors (KAB) survey |

#### ATTACHMENTS:

Original protocol: 'LRTIR01protocol.12 23 2013'

Data collection protocols and forms: 'Child Health Measures Visit Protocol 10272014'

End of Winter Home Questionnaires and KAB survey: 'End of Winter Questionnaires and KAB 11112015'

Statistical Analysis Plan

Form RA-108 (Rev. 11/13)

#### THE UNIVERSITY OF MONTANA-MISSOULA

Institutional Review Board (IRB)
for the Protection of Human Subjects in Research
CHECKLIST / APPLICATION

| IRE | 3 Pro | otoc | col | No. | : |
|-----|-------|------|-----|-----|---|
| | | | | | _ |

At the University of Montana (UM), the Institutional Review Board (IRB) is the institutional review body responsible for oversight of all research activities involving human subjects outlined in the U.S. Department of Health and Human Services' Office of Human Research Protection and the National Institutes of Health, Inclusion of Children Policy Implementation.

**Instructions:** A separate application form must be submitted for each project. IRB proposals are approved for no longer than one year and must be continued annually (unless Exempt). Faculty and students may email the completed form as a Word document to <a href="IRB@umontana.edu">IRB@umontana.edu</a>. or submit a hardcopy to the Office of the Vice President for Research & Creative Scholarship, University Hall 116. Student applications must be accompanied by email authorization by the supervising faculty member or a signed hard copy. *All fields must be completed. If an item does not apply to this project, write in: n/a.* Questions? Call 243-6672.

| Project Title: Wood stove interventions and child respiratory infections | | | | | | | |
|---|---|---|---|---|---|---|---|
| Principal Investigator: Curtis Noonan and Tony Ward | | | | UM Position: Assoc Professor | | | |
| | EHS/BMED | | | | Office location: S | Skaggs | |
| Work Phone: 4 | 06-243-4957 | | | | Cell Phone: | | |
| study course on | ojects Protection Training<br>protection of human research s<br>Certificate(s) of Completion" up | ubjects <b>within t</b> | he last three | e years ( <u>ht</u> i | <u>p://www.umt.ed</u> | <u>u/research/co</u> | omplianceinfo/IRB/) and |
| | esearch Team Members (list yourse | | PI | СО-РІ | Faculty | Research<br>Assistant | DATE COMPLETED Human Subjects Protection Course |
| Name: Curtis | Noonan | | $\boxtimes$ | | | | 9/20/2011 |
| | noonan@umontana.edu | | | | | | |
| Name: Tony | | | | | | | 12/28/2012 |
| | vard@umontana.edu | | | | | | |
| Name: Erin S | | | | | | | 3/26/2013 |
| | emmens@umontana.edu | | | | | | |
| Name: Desira | | | | | | $\boxtimes$ | 11/4/2013 |
| Email: desira | e.ware@umontana.edu | | | | | | |
| agency? X Agency NIEHS | Yes (If yes, cite sponsor on ICI Grant No. | F if applicable) Start | | | s <i>(If yes, cite spo</i><br>End Date | P | <i>if applicable)</i> ⊠No I on grant Vard and Noonan |
| | | I | | | | | |
| _ Not Huma<br>_ Approved | ermination: an Subjects Research by Exempt Review, Cate by Expedited Review, Ca | | · | )<br>te to PI) | only. Use any at<br>as "masters" who<br>the expiration da<br>Notify the IRB i<br>events occur. We<br>must be submitted | ttached IRB-<br>en preparing<br>ite, a continu<br>f any signific<br>then the stud | dies are approved for on<br>approved forms (signed/<br>copies. If continuing be<br>ation report must be sub-<br>cant changes or unanticip<br>y is completed, a closure<br>follow these directions |
| | Determination | | · | | constitutes non-c | | vitii OWi policy. |
| Full IRB | Determination proved (see Note to PI) | | | | constitutes non-c | Р | with OW policy. |
| Full IRB <br>Ap<br>Co | Determination proved (see Note to PI) nditional Approval (see me Conditions Met (see No | mo) - IRB Cha<br>ote to PI) | ir Signature | /Date: | | | |
| Full IRB Ap | Determination proved (see Note to PI) nditional Approval (see me | mo) - IRB Cha<br>ote to PI) | ir Signature/ | /Date: | | | vitii Oivi policy. |

<In an effort to be environmentally responsible, please expand/reduce box size as needed.>

4. Purpose of the Research Project: Briefly summarize the overall intent of the study. Your target audience is a non-researcher. Include in your description a statement of the objectives and the potential benefit to the study subjects and/or the advancement of your field. Generally included are literature related to the problem, hypotheses, and discussion of the problem's importance. Expand box as needed.

Acute lower respiratory tract infections (LRTIs) account for more than 27% of all hospitalizations among US children under five years of age, with recurrent LRTIs in children a recognized risk factor for asthma. Within rural areas of Montana, Alaska, and the Navajo Reservation, research has shown that residential biomass combustion leads to elevated indoor levels of fine particulate matter (PM2.5) that often exceed current healthbased air quality standards. Parallel findings have been observed in several developing countries where biomass combustion is commonly used for cooking and/or heating. This is concerning, as PM2.5 exposure is associated with many adverse health outcomes, including a greater than three-fold increased risk of LRTIs. Currently, there is a global effort to reduce indoor biomass smoke exposures in developing countries through the introduction of improved cookstove technology. Similar evidence-based efforts are warranted in rural and Native American communities in the US that suffer from elevated rates of childhood LRTI and commonly use wood for residential heating. To date, exposure reduction strategies in wood stove homes have been either inconsistently effective or include factors that limit widespread dissemination and continued compliance in rural and economically disadvantaged populations. In this project, we propose to test the efficacy of two intervention strategies for reducing indoor wood smoke PM2.5 exposures and children's risk of LRTI in three unique and underserved settings: (1) rural mountain valley communities in western Montana; (2) Navajo Nation communities; and (3) Alaska Native Villages. We will conduct a three-arm randomized placebo-controlled postonly intervention trial in wood stove homes with children less than five years old. Education on best-burn practices and training on the use of simple instruments (i.e., stove thermometers and wood moisture meters) will be introduced as one intervention arm (Tx1). This intervention will be evaluated against an indoor air filtration unit arm (Tx2), as well as a placebo arm (Tx3, sham air filters). The primary outcome will be LRTI incidence among children under five years of age. To allow for detection of exposure and outcome differences within each of the three regions, a sample of 324 homes, or 108 within each study area will be equally assigned to each of the three intervention arms. The overall hypothesis is that a low-cost, educational intervention targeting indoor wood smoke PM2.5 exposures will be sustainable, and can reduce children's risk of LRTI in underserved Native and rural communities.

This checklist submitted to the University of Montana IRB is specific for the activities in study area 1: rural mountain valley communities in western Montana. As indicated below (item #5) the other two study sites will fall under the jurisdication of the respective local IRBs.

| 4.1 | What do you plan to do with the results? If not discussed above, include considerations such as whether this is a class project, a |
|---|---|
| proje | ect to improve a program/school system, and/or if the results will be generalized to a larger population, contribute to the general field |
| of kn | nowledge, and/or be published/presented in any capacity. |

| | Results will be generalized to other communities and households that burn biomass for residential heating. Results of this research will be published in peer reviewer journals. |
|---|---|
| | Is this part of a thesis or dissertation? \( \sum No \) \( \sum Yes \) If yes and other than the PI's, then whose? |
| 5. II | IRB Oversight Is oversight required by other IRB(s) [e.g., tribal, hospital, other university] for this project? ☑ Yes ☐ No If yes, please identify IRB(s): |
| | This study will be approved by The University of Montana Institutional Review Board (UM-IRB). Approval for study site 2 will be submitted to the Navajo Nation Human Research Review Board. Approval for study site 3 will be submitted to the Alaska Area Institutional Review Board (AAIRB), and the Yukon Kuskokwim Health Corporation Human Studies Committee. |

#### 6. Subject Information:

6.1 Human Subjects (identify, include age/gender):

Eligible subjects will include children less than 5 years of age that live in a household that utilizes a wood stove as the primary heating source in the study region (i.e., rural Montana). We anticipate an equal number of male and female child participants. A total of 108 households from this study area will be recruited for this study. We assume approximately 1.5 children under 5 years old per household (n = 162 total child subject).

| 6.2 How many subjects will be included in the study? <u>162</u> |
|---|
| 6.3 Are minors included (under age 18, per Montana law)? ☐ Yes ☐ No If yes, specify age range: 0 to 5 |
| 6.4 Are members of a physically, psychologically, or socially vulnerable population being specifically targeted? Yes No |
| If yes, please explain why the subjects might be physically, psychologically or socially vulnerable: |
| 6.5 Are there other special considerations regarding this population? Yes No If yes, please explain: |
| 6.6 Do subjects reside in a foreign country? Yes Specify country: No If yes, please fill out and attach Form RA-112, Foreign Site Study Appendix (http://www.umt.edu/research/complianceinfo/IRB/Docs/foreign.doc). |
| 6.7 How are subjects selected or recruited? Include a bulleted list of inclusion/exclusion criteria. (Attach copies of all flyers, advertisements, etc., that will be used in the recruitment process as these require UM-IRB approval) For the western Montana study area, we will recruit participants through the local medical center, pediatricians' offices, and the Women, Infants and Children (WIC) programs. In addition, we will communicate directly with obstetricians, pediatricians, and WIC community nurses to describe the study, and provide recruitment materials such as flyers and post cards to be returned by potentially eligible participants. |
| Inclusion criteria: - Eligible homes will be any home that uses a wood stove as a primary heating source, and has one or more children under the age of five years. The home must include a parent who is capable and willing to record symptom data for the enrolled children and wood stove usage data. Exclusion criteria: |
| - None. |
| 6.8 How will subjects be identified in your personal notes, work papers, or publications: (may check more than one) [ Identified by name and/or address or other (Secure written [e.g., ICF] or verbal permission to identify; if risk exists, create a confidentiality plan.) |
| ☑ Confidentiality Plan (Identity of subjects linked to research, but not specific data [e.g., individuals identified in ICF but not included it publications]; identification key kept separate from data; or, data collected by third party [e.g., Select Survey, SurveyMonkey, etc.] and identifiers not received with data.) |
| Never know participant's identity (An ICF may be unnecessary [e.g, anonymous survey, paper or online] unless project is sensitive or involves a vulnerable population.) |
| 6.9 Describe the means by which the human subject's personal privacy is to be protected, and the confidentiality of information maintained. If you are using a Confidentiality Plan (as checked above), include in your description a plan for the destruction of materials that could allow identification of individual subjects or the justification for preserving identifiers. |
| All households, and child subjects within household, will be assigned unique identification numbers. For practical purposes, the PI or appropriate study personnel will have a linkage file on-site (e.g., a file that identifies the subjects and their corresponding numbers) during the data collection days to ensure that the correct subjects are identified. At all other times, this linkage file will be under the control of the University of Montana PIs. The linkage file will be kept separate from other data materials. When sample collection is completed, this linkage file will be returned to a locked file cabinet under the control of Co-PI Noonan. Data will be recorded on data collection sheets that contain only the subject's identification number and no other personal identifiers. |

| | 6.9a Will subject(s) receive an explanation of the research – separate from the informed consent form (if applicable) – before and/or after the project? Yes (attach copy and explain when given) No |
|---|---|
| 7. | Information to be Compiled |
| | 7.1 Explain where the study will take place (physical location not geographic). If permission is required to conduct the research at the location or to use any of the facilities, indicate those arrangements and attach copies of written permission |
| | The study will take place in the children's homes. |
| | 7.2 Will you be working with infectious materials, ionizing radiation, or hazardous materials? Please specify. |
| | N/A |

#### 7.3 Subject matter or kind(s) of information to be compiled from/about subjects:

The primary health outcome will be occurrence of LRTI among children, and will be assessed using active surveillance within the home. Identification of LRTI episodes will occur through a three step process: (1) parent reporting of symptoms; (2) Community Coordinator collection of confirmatory and severity data; and (3) physician classification of case status based on data collected by the Community Coordinator, and when available, data collected from a clinic or hospital.

At the onset of the program in each study area, comprehensive health outcomes assessment training of Community Coordinators will be provided by Drs. Paul Smith and Curtis Noonan, Community Coordinators will then train parents in the identification of symptoms consistent with LRTI (cough, difficulty breathing, fast breathing, noisy breathing, nasal discharge, loss of appetite and fever). Parents will be asked to contact their Community Coordinator when such symptoms are present in household children < five years (Step 1). Home visits will occur within 48 hours of parent notification of signs and symptoms of LRTI. At this visit, the Community Coordinator will interview the parent about each study participant's symptoms. The Community Coordinator will then measure temperature, respiratory rate and saturated oxygen, and evaluate the child for presence of chest indrawing (retractions), wheeze and cough (Step 2). Please note that the Community Coordinators are not diagnosing respiratory illness or providing medical care, and parents will be encouraged to seek medical care for treatment of their child's respiratory symptoms, when indicated (see also Protection of Human Subjects section). For any study participant experiencing symptoms, the Community Coordinator will document the presence of symptoms and date of onset with the parent. During the regular communication with the parent and subsequent home visits, the Community Coordinator will continue to track this child's symptoms. The last day of cough and rapid breathing with no recurrence of symptoms during a following 14 day period will be considered the end date for a given episode. Per approaches used internationally, if symptoms recur within a period of less than 14 days, these symptom days will be considered part of the immediately preceding episode rather than a separate episode. Days with cough as the only symptom will not be included as days for the given LRTI episode. The Community Coordinator will also determine if the child was observed by a health care provider, clinic or hospital during this episode. If available, health data from such visits will be collected from the covered entity with the corresponding parent-signed HIPPA forms. Data collected from medical records will include health care provider diagnosis, ausculatory findings, and laboratory/radiological findings.

The Step 1 strategy may be adversely impacted by lack of follow-up by the parent or communication barriers that may vary by community. To address this, the Community Coordinator will engage in active and frequent surveillance of homes (Step 2), interviewing the parent at a minimum of once every two weeks regarding symptoms among study participants. This communication will occur via telephone, email, or a home visit depending upon the community setting and the preferred method of communication. The Community Coordinator will also visit the home at a minimum of once per month to measure respiratory rate and saturated oxygen, regardless of whether or not the parent has reported child symptoms consistent with LRTI. When indicated the Community Coordinator will collect objective measures and prospectively track symptoms according to the Step 1 procedures indicated above.

For primary analysis, the final case determination will be made by pediatric pulmonologist, Paul Smith, D.O (Step 3). The primary case definition will be based on the objective data collected by the Community Coordinator. Children <5 years will be considered to have LRTI if the Community Coordinator documents cough and a respiratory rate ≥40 breaths per minute in children <1 year or ≥30 breaths per minute in children 1 to <5 years. The primary determinants of LRTI status (i.e., respiratory rate and presence of cough) are easily captured by trained Community Coordinators. The respiratory rate thresholds are highly sensitive indicators for presence of LRTI. To improve specificity for LRTI, Dr. Smith will further distinguish between moderate and severe LRTI (i.e., secondary case status determination)

according to the presence of fever, chest indrawing, wheeze and saturated oxygen readings <90% as documented from direct field observation or from clinical records.

Other data collection: We will capture additional data that may be relevant to either risk of LRTI or PM2.5 exposures. Individual-level characteristics to be captured from parents will include child's vaccination history, occurrence and duration of breastfeeding, birth weight, and maternal age. Household-level characteristics will include crowding, presence of mold, cleanliness, parent education level, household income, and household tobacco smokers. To supplement the reporting of household tobacco use, we will collect household surface dust wipe samples at each exposure sampling visit to measure deposited nicotine. Alcohol wipes will be collected from horizontal surface areas within the home in areas that are not frequently cleaned (top of doors, top of cabinets, etc.). Following a revised method utilized by the US Centers for Disease Control and Prevention,101 analysis for nicotine will be performed from the wipes using Gas Chromatography/Mass Spectrometry (GC/MS) at UM under the direction of Dr. Tony Ward. Exposures could also be impacted at the household level by various factors such as the use of power generators or the use of materials other than wood in stoves, with some activities specific to the study sites.

7.4 Activities the subjects will perform and how the subjects will be used. Describe the instrumentation and procedures to be used and kinds of data or information to be gathered. **Provide enough detail** so the IRB will be able to evaluate the intrusion from the subject's perspective (expand box as needed):

During assessment of suspected LRTI, the Community Coordinator will measure the child's temperature, respiratory rate and saturated oxygen, and evaluate the child for presence of chest indrawing (retractions), wheeze and cough. This will take approximately 15 minutes for each time these factors are assessed for a given child. These same measures will be captured for the child each time the Community Coordinator visits the child's home. These visits will occur once per month for two six-month winter periods, or a total of 12 visits.

| 7.5 | Is information on any of the following included? (check a Sexual behavior Alcohol use/abuse Information about the subject that, if it became kn subject at risk of criminal or civil liability or be deemployability. | Drug use/abuse Illegal conduct nown outside the research, could reasonably place the |
|---|---|---|
| 7.6 | Means of obtaining the information (check all that apply). | Attach questionnaire or survey instrument, if used: |
| | ☐ Field/Laboratory observation | In-person interviews/survey |
| | Blood/Tissue/Urine/Feces/Semen/Saliva | Telephone interviews/survey |
| | Sampling (IBC Application must be submitted) | On-site survey |
| | ✓ Medical records (require HIPAA form) | Mail survey |
| | Measurement of motions/actions ■ Me | Online survey (attach Statement of Confidentiality) |
| | Use of standard educational tests, etc. | Examine public documents, records, data, etc. |
| | Other means (specify): | Examine private documents, records, data, etc. |
| 7.7 | Will subjects be (check all that apply): | |
| | ☐ Videotaped ☐ Audio-taped | ☐ Photographed ☐ N/A |
| | (securing an additional signature is recommo | ended on consent/assent/permission forms) |
| | Explain how above media will be used, who will trans | |
| | | · |

7.8 Discuss the benefits (does not include payment for participation) of the research, if any, to the human subjects and to scientific knowledge (if the subjects will not benefit from their participation, so state):

Those who participate in this research may help inform health researchers, physicians, and the regulatory community about exposure to smoke from wood stoves and the impact of these exposures on susceptible populations. These findings will help identify interventions that will be generalizable to other rural impacted by wood smoke. Information collected from exposure assessments will also be made available to subjects at the end of their participation in the study. These data could be useful for identifying strategies to mitigate in home exposures to PM and respiratory morbidity among children. The study may benefit study participants directly through the collection of objective measures of their respiratory health. Although the Community Coordinators will not be diagnosing children or providing them with medical care, they will have information on normal ranges for respiratory rate, oxygen saturation, temperature and retractions and thus can refer children for medical care or make a recommendation for referral. In these cases, the participants may benefit from receiving care that they might not otherwise have sought.

7.9 Cite any payment for participation (payment is not considered a benefit). If grant funding is not indicated in item #2, please specify the source of the funding and in what form it is to be dispersed.

Households, rather than the child subjects, will be payed for their participation. Each household participating in the project in western Montana will receive \$100 per each of two winter periods, or a total of \$200.

7.9a Outline, **in detail**, the risks and discomforts, if any, to which the human subjects will be exposed (Such deleterious effects may be physical, psychological, professional, financial, legal, spiritual, or cultural. As a result, one can never guarantee that there are no risks – use "minimal." Some research involves violations of normal expectations, rather than risks or discomforts; such violations, if any, should be specified):

This study will be conducted in the home of children less than 5 years of age. The household intervention does not involve any medications or changes to the child's normal care. The proposed methods for assessing the presence of LRTI are non-invasive, including respiratory rate measures and recording of symptoms.

7.9b Describe, in detail, the means taken to minimize each such deleterious effect or violation::

The Coordinators will be trained by our medical consultant to recognize when a child's symptoms indicate the need for medical referral.

#### 8. Informed Consent

An informed consent form (ICF) is usually required, unless subjects remain anonymous or a waiver is otherwise justified below. (Templates and examples of Informed Consent, Parental Permission, and Child's Assent Forms are available at <a href="http://www.umt.edu/research/complianceinfo/irb/forms.aspx">http://www.umt.edu/research/complianceinfo/irb/forms.aspx</a>).

- A signed copy of the consent/assent/permission form must be offered to all subjects, including parents/guardians of subjects less than 18 years of age (minors).
- Use of minors
  - All minor subjects (under the age of 18) must have written parental or custodial permission (45 CFR 46.116(b)).
  - o All minors from 10 to 18 years of age are required to give written assent (45 CFR 46.408(a)).
  - Assent by minor subjects: All minor subjects are to be given a clear and complete picture of the research they are being asked to engage in, together with its attendant risks and benefits, as their developmental status and competence will allow them to understand.
  - Minors less than 10 years of age and all individuals, regardless of age, with delayed cognitive functioning (or with communication skills that make expressive responses unreliable) will be denied involvement in any research that does not provide a benefit/risk advantage.
    - Good faith efforts must be made to assess the actual level of competence of minor subjects where there is doubt.
    - The Minor Assent Form must be written at a level that can be understood by the minor, and/or read to them at an age-appropriate level in order to secure verbal assent.

| • | Is a written informed consent form being used? Yes (attach copy) No (justify below) |
|---|---|
| | To waive the requirement for written informed consent (45 CFR 46.117), describe your justification: |
| | <u>_</u> |
| • | Is a written parental permission form being used? \( \sum \text{Yes (attach copy)} \sum \subseteq \text{No} \) |
| | (If yes, will likely require minor assent form) |
| • | Is a written minor assent form being used? \( \sum \text{ Yes (attach copy)} \sum \text{No} \) |
| | (If yes, will likely require parental permission form) |

#### Principal Investigator's Statement

By signing below, the Principal Investigator agrees to comply with all requirements of The University of Montana-Missoula IRB, the U.S. Department of Health and Human Services Office of Human Research Protection Guidelines, and NIH Guidelines. The PI agrees to ensure all members of his/her team are familiar with the requirements and risks of this project, and will complete the Human Subject Protection Course available at <a href="http://www.umt.edu/research/complianceinfo/irb">http://www.umt.edu/research/complianceinfo/irb</a>.

I certify that the statements made in this application are accurate and complete. I also agree to the following:

• I will <u>not</u> begin work on the procedures described in this protocol, including any subject recruitment or data collection, until I receive <u>final</u> notice of approval from the IRB.

- I agree to inform the IRB in writing of any adverse or unanticipated problems using the appropriate form. I further agree not to proceed with the project until the problems have been resolved.
- I will not make any changes to the protocol written herein without first submitting a written **Amendment Request** to the IRB using form RA-110, and I will not undertake such changes until the IRB has reviewed and approved them.
- It is my responsibility to ensure that every person working with the human subjects is appropriately trained.
- All consent forms and recruitment flyers must be approved and date-stamped by the IRB before they can be used. The
  forms will be provided back to the PI in PDF format with the IRB approval email. Copies must be made from the datestamped version. All consent forms given to subjects must display the IRB approval date-stamp.
- I understand that it is <u>my responsibility</u> to file a **Continuation Report** before the project expiration date (does not apply to exempt projects). This is not the responsibility of the IRB office. *Tip: Set a reminder on your calendar as soon as you receive the date.* A project that has expired is no longer in compliance with UM or federal policy.
- I understand that I must file a **Closure Report** (RA-109) when the project is completed, abandoned, or otherwise qualifies for closure from continuing IRB review (does not apply to exempt projects).
- I will keep a copy of this protocol (including all consent forms, questionnaires, and recruitment flyers) and all subsequent correspondence with the IRB.
- I understand that failure to comply with UM and federal policy, including failure to promptly respond to IRB requests, constitutes **non-compliance** and may have serious consequences impacting my project and my standing at The University of Montana.

| Signature of Principal Investigator: | Date: | |
|---|---|---|
| | Type for electronic submission; sign for hard copy) | _ |
| NOTE: I AM AWARE that electro | ic submission of this form from my University email account constitutes my signature | €. |
| <b>Students and Faculty Advisors:</b> S supervising faculty member or by a | udent applications must be accompanied by either an email authorization from the igned hard copy (below). | |
| Faculty Supervisor: | | |
| 2) I agree that it ac | RB Application and attachments. surately represents the planned research. this research project. | |
| Faculty Advisor Signature: (Type for e | Date: ectronic submission; sign for hard copy) | |
| Department: | Phone: | |

#### **Child Health Measures Contacts and Visits**

#### *Initial visit (at time of recruitment/informed consent):*

- 1. Review parental permission form and answer parent questions.
- 2. Review and complete HIPAA form.
- 3. Obtain assent from children age 4 and 5 years of age
- 4. Upon the receipt of signed parental permission (for all children) and child assent (for children ages 4-5 years), study personnel will ask the contact parent to complete the following documents:
  - A. Demographics Form
  - B. <u>Home Characteristics Form</u>
  - C. Child Birth and Infancy Data
  - D. <u>Authorization to Use and Disclose Protected Health Information for Research Purposes</u>

#### Phone contacts and procedures for parent-reporting of child symptoms:

- Provide study phone numbers.
- Provide instruction sheet for identifying child symptoms (see <u>PARENT/CAREGIVER</u> REPORTING OF SYMPTOMS).
- When parent contacts study personnel, <u>Child Symptom Questionnaire</u> (below) will be completed.

Study personnel also will monitor child symptoms via phone call with contact parent at a frequency of once per two weeks during the winter period. Home visits will supersede phone-based data collection.

In phone communications, the <u>Child Symptom Questionnaire</u> will be completed.

#### Home visits and data collections:

Home visits will occur at a frequency of once per month during the winter period, or as indicated by phone contact that was initiated either by study personnel or contact parent.

Note: Even if the visit is initiated by illness report for a given child, when another study child resides in the same home, these data also will be collected for that symptom-free child.

At home visit, the following will be collected for each child participant:

- <u>Child Symptom Questionnaire</u> (parent response)
   Note: Even if these symptom data were collected during a phone contact, these symptom data should be collected again at home visit.
- <u>Health Measures Visit Sheet</u>. Protocols for the following are included:
  - Respiratory rate
  - Heart rate and saturated oxygen (i.e., pulse oximetry)
  - Temperature

See also Referral Protocol.

#### Capture of data from child's health provider visit, when applicable:

If the parent has indicated that the child has been taken to a health care provider (see Child Symptom Questionnaire), study personnel will request data from the respective health care provider. Per the parent-signed "Authorization to Use and Disclose Protected Health Information for Research Purposes," the following data will be requested:

- Diagnosis of respiratory tract infection, including both upper and lower respiratory infection;
- Lab results related to respiratory tract infection
  Any results from respiratory "swabs" if obtained (RSV, influenza, pertussis, parainfluenza)
- presence of fever;
- observation of chest retractions;
- wheeze or other impaired breathing symptoms; and
- saturated oxygen readings
- chest radiographic information (positive or negative findings)

#### **Exposure sampling visits:**

During the first winter, up to two sampling visits will occur to collect indoor air quality data. The air sampling equipment will be placed by study personnel and will measure temperature and dust for up to 6 days. The home participants will not need to assist with the air sampling equipment, but we will ask them to complete the following forms:

- Home characteristics
- Home activity Log
- Wood stove usage
- In-home Log

| <b>Demographic Questions for Primary Caregiver</b> | | | Home ID: |
|---|---|---|---|
| | | | Date: |
| 1. | Please circle one: | Female | Male |
| 2. | Are you Hispanic or Latir | Are you Hispanic or Latino? | |
| | Yes | No | |
| 3. | What is your race? Circle | e one or more races to | indicate what you consider yourself to be: |
| | American Indian/ | Alaskan Native | |
| | Asian | | |
| | Native Hawaiian | or Other Pacific Islande | er |
| | Black or African A | American | |
| | White | | |
| | More than one rad | ce | |
| 4. | Circle the category that b | est describes your hou | usehold income? |
| | Less than \$20,00 | 0 | |
| | \$20,000 to \$29,99 | 99 | |
| | \$30,000 to \$39,99 | 99 | |
| | \$40,000 to \$49,99 | 99 | |
| | \$50,000 to \$74,9 | 99 | |
| | \$75,000 to \$99,9 | 99 | |
| | \$100,000 or more | e | |
| 5. ( | Circle the category that be | est describes your year | rs of school completed: |
| | Less than high so | chool | |
| | High school diplo | ma or GED | |
| | Some college | | |
| | College degree | | |
| 6. | How many total residents | s are in your home? | |
| 7. | How many children unde | er 5 reside in your home | e? |

# If you have more than one child under 5 years of age, please answer the following questions starting with the youngest child first:

| Qι | estions for Child #1 | | | |
|---|---|---|---|---|
| 8. | 3. Is your child Hispanic or Latino? | | Age of Child # | 1 on November 1st: |
| | Yes | No | | |
| 9. | What race is your child? | | | |
| | American Indian | /Alaskan Native | | Asian |
| | Native Hawaiian | or Other Pacific | Islander | Black or African American |
| | White | | | More than one race |
| Qι | estions for Child #2 | | | |
| 10 | . Is your child Hispani | c or Latino? | Age of Child #2 | 2 on November 1st: |
| | Yes | No | | |
| 11 | . What race is your ch | ild? | | |
| | American Indian | /Alaskan Native | | Asian |
| | Native Hawaiian | or Other Pacific | Islander | Black or African American |
| | White | | | More than one race |
| Qι | estions for Child #3 | | | |
| 12 | . Is your child Hispani | c or Latino? | Age of Child #3 | on November 1st: |
| | Yes | No | | |
| 13 | . What race is your ch | ild? | | |
| | American Indian/Alaskan Native | | | Asian |
| | Native Hawaiian | or Other Pacific | Islander | Black or African American |
| White | | | | More than one race |

# HOME CHARACTERISTICS DATA SHEET

| Technician: | Home ID: | Winte | er (1,2,3, | etc.): |
|---|---|---|---|---|
| Sampling Dates: | Date form co | ompleted: | | |
| To be completed by an ac | dult resident on | ce at the begi | nning | of each winter. |
| 1. Number of total residents in | n home: | | | |
| 2. Number of residents young | er than 18 years of | age: | | |
| 3. Number of residents young | er than 5 years of a | .ge: | | |
| 4. Type of home: House | Mobile Home | Duplex/Apt | Other: | |
| 5. Year home built: | | | | |
| 6. Square footage of home: | | | | |
| 7. Number of floors (not incl. | bsmnt): 1 | 2 3 | | |
| 8. Number of windows: | | | | |
| 9. Number of bedrooms: | | | | |
| 10. Total number of pets: | | | | |
| 11. Total number of "furry" pe | ts: | | | |
| 12. Type of primary heating (P | lease circle ONLY | one choice that | represei | nts your most common practice): |
| Wood stove Electrical | Propane Natu | ıral gas furnace | Oil | Other: |
| 13. Type of secondary heating | (Please circle <b>ONL</b> | Y one choice th | at repres | sents your most common practice): |
| Wood stove Electrical | Propane Natu | ıral gas furnace | Oil | Other: |
| 14. Existing appliance(s): Fire | eplace Wood stor | ve Furnace | Wood | stove insert |
| 15. Wood stove model (If you i | have access, inform | nation is located | on the b | pack of the stove): |
| 16. Approximately how old is | your wood stove: | | | |
| 0-5 years old 6-10 years | ars old 11-1 | 5 years old | 16 + v | ears old |

| 17. | Is your wood | l stove EPA- | certified? | Yes | No | I don' | t know |
|---|---|---|---|---|---|---|---|
| 18. | When was th | e last time y | ou had your | chimney c | leaned? | | |
| | Less than 6 n | nonths ago | 6-12 mor | nths ago | 12-18 month | ns ago | more than 18 months ago |
| 19. | | | - | | lamp spots on<br>lings or carpet | | s inside your home other than in the |
| | Yes | No | I don't kno | w | | | |
| 20. | Has there bee | en mold or n | nildew on ar | y surfaces | inside your ho | ome in t | he last 12 months? |
| | Yes | No | I don't kno | W | | | |

# **Child Birth and Infancy Data** Technician: Home ID #: \_\_\_\_\_ Child ID #:\_\_\_\_\_ Date of Birth: Age: Sex: Birth weight: \_\_\_\_\_ Age of Mother at Birth: Breastfed? (circle one) Yes No If yes, for how long? Has your child received the flu shot this year? (circle one) No Yes If not, do you plan to have your child receive the flu shot? Yes No

Does your child attend: day care preschool/school

If yes, how many hours/day: \_\_\_\_\_ How many days/week: \_\_\_\_\_

Does your child have siblings in school or day care? Yes No

#### PARENT/CAREGIVER REPORTING OF SYMPTOMS - INSTRUCTIONS

We are asking you to help us in monitoring the health of your child. We would like you to contact us immediately if your child experiences any of the symptoms indicated below.

You can contact us through one of two ways:

- 1. By email to KidsAIR@umontana.edu.
- 2. By voice message or text to 406-?????

As part of your email, voice or text message please indicate a good time for us to call you back on that day or the next.

#### PLEASE NOTIFY US IF YOUR CHILD EXPERIENCES ANY OF THE FOLLOWING:

- Fever
- Rapid breathing
- Difficult breathing
- Noisy breathing
- Runny nose
- Cough
- Wheezing
- Doctor or health clinic visit for any of the above

Procedures for collection of child health measures (i.e., respiratory rate, saturated oxygen, temperature). Complete the Child Symptom Questionnaire and Health Measures Visit Sheet.

- 1. Make sure the child is comfortable with who you are and what you intend to do.
- 2. Explain your steps to them beforehand so they are aware.
- 3. Very young children may want to play with or touch your equipment as well, and it will most likely calm them if they do. Both instruments are rugged and can withstand being handled by them.

#### **History/Symptoms**

- 4. Make sure you have your Child Symptom Questionnaire handy for recording data.
- 5. Complete the questionnaire and record symptoms as stated by the caregiver. You can also make note of symptoms given by the child if they offer them up (but write them separately so you know which comments belong to whom). Record any important personal observations as well.

#### **Health Measures**

- 6. Per training with Dr. Paul Smith, complete the Health Measures Visit Sheet.
- 7. Count and observe respiratory rate and effort. It is best if the caregiver can hold the child on their lap with their shirt up. She can distract or comfort them while you observe. Determining respiratory rate can be easy if the child is distracted by something (like a toy or TV), or if the child is sleeping. With older children, or very attentive ones, it can be harder to observe their breathing rate without them noticing. If the child knows you are counting their breaths, they may adjust their breathing rate subconsciously. A good trick is to instead act like you are taking their pulse, and while they think you are feeling for their heartbeat at the wrist, you are instead subtly watching them inhale and exhale. You can also place a hand flat on the child's upper back to help feel inhalations and exhalations better.
  - When counting breaths, you will need to have a clock nearby.
  - Start counting breaths for 30 seconds and remember the number.
  - Take this number and multiply it by 2. This is the number of breaths per minute.
  - Record this observation in the Health Measures Visit Sheet.
  - Also note any retractions in the Health Measures Visit Sheet.
- 8. Now, take the child's temperature using the temporal thermometer. This thermometer simply touches their forehead, and is very noninvasive. See the <a href="EXERGEN Temporal Thermometer">EXERGEN Temporal Thermometer</a> Protocol.
- 9. Chest auscultation for crackles, wheeze or stridor.
- 10. Determine the Oxygen saturation (SpO2) in the blood by using the Pulse Oximeter next. See the <u>Pulse Oximeter Protocol</u>. Do this last. Some kids hate it and crying will make the rest of your exam hard. Also record the pulse rate (PRbpm) off the SpO2.

## **CHILD SYMPTOM QUESTIONNAIRE**

| Home ID # | | Child ID # | | | | |
|---|---|---|---|---|---|---|
| Date: | | Data collected: | By phone | At home | | |
| In the last two | o weeks has your ch | ild been ill? | | No | Yes | |
| If yes, is child | still ill? | | | No | Yes | |
| Has your child | d seen a doctor or h | ospital or nurse for | this illness? | No | Yes | |
| • | e person/location:_<br>ider is different fror<br>rm. | n indicated on PHI | form collected a | t initial visit, o | obtain a new par | ent |
| Is your child t | aking any new med | icines for this illnes | ss? | No | Yes | |
| Medication N | ames | | | | | |
| | d had any of the foll | owing: | | | | |
| | Fever? | | No | Yes | | |
| | | | | • | perature?<br>N/A" if unknown. | |
| | Rapid breathing? | | No | Yes | | |
| | Difficult breathin | g? | No | Yes | | |
| | Noisy breathing? | | No | Yes | | |
| | Runny nose? | | No | Yes | | |
| | Cough? | | No | Yes | | |
| | Wheezing? | | No | Yes | | |

[If data were collected by phone and child is currently ill, schedule home visit]

| <b>Health Measures</b> | Visit Sheet |
|------------------------|-------------|
|------------------------|-------------|

| Home ID # | Child ID # |
|-----------|------------|
| Date: | |

### **Physical**

| Lethargy | RR | Retractions | Temperature °F | Lung sounds | %SpO2 | Heart Rate | AHR |
|---|---|---|---|---|---|---|---|
| Vas. Na | (bpm) | (score) | | Wheeze | | (PRbpm) | |
| Yes No | | | | Stridor | | | |
| | | | | Crackles | | | |

Referred? Yes No If yes, indicate level of referral: Emergent Urgent Recommended follow up with primary care provider

**Note:** For an Emergent or Urgent referral, follow referral procedures and then contact PI immediately.

#### **EXERGEN Temporal Thermometer Protocol**

- 1. Remove cap from the end of thermometer.
- 2. Make sure metal probe surface is shiny and clean.
  - a. If not, use an alcohol swab to clean.
  - b. Allow to dry.
- 3. Place probe end of thermometer flush to the center of child's forehead.
  - a. Probe should be halfway between hairline and eyebrows.
- 4. With the probe placed, press the grey front button and hold.
  - a. The thermometer will start beeping and a red LED on the back of the thermometer will turn on.
- 5. With the button still depressed, slide the thermometer from the center of the forehead left or right to the hairline.
  - a. Keep the probe moving in a straight line—don't follow the hairline down toward the ear.
- 6. Release the grey button when you reach the hairline.
- 7. Your temperature measurement will show on the LED display.
- 8. Record temperature on Health Measures Visit Sheet.
- 9. Clean probe sensor area with an alcohol swab.
- 10. Allow to dry and reattach probe cap for travel.
- 11. To switch the battery, remove the back lower cover and exchange the 9V square battery.





The thermometer will turn off on its own. To wake it back up, press the grey button once. The display will then show you the last measurement taken. If you continue to hit the grey button, it will scroll through the last eight measurements taken.

### \*If the forehead has perspiration present, measure the temperature from behind the ear instead.

- 1. Instead of placing probe on center of forehead, place it on the neck just behind the ear lobe.
- 2. Press and hold grey button as before and take a reading while keeping the probe stationary in that spot.





#### **Pulse Oximeter Protocol**

- 1. Remove blue Pulse Oximeter (pulse-ox) from blue carrying case.
- 2. Squeeze the end of the pulse-ox that says PUSH to open the clip.
- 3. Place the child's index or thumb into the clip and release the pulse-ox so it gently squeezes the finger.
  - a. The child's fingernail should be facing up, toward the display. Don't put the pulse-ox on upside down!
  - b. Make sure the child is not moving and is at ease during this process.
- 4. Press the white button on the top and it will turn on and start to take a reading.
  - a. You'll notice red LED lights show up on the display.
  - b. The reading will take a few seconds before it shows up on the display.
  - c. Once it's ready, you will see two numbers:
    - i. The first number will appear about "PRbpm," which is your current Heart Rate
    - ii. The second number appears above "%SpO2," which is your oxygen percentage.
  - d. Wait at least 10 seconds after the first reading shows up before you record the numbers.
  - e. Write the two measurements down on the Health Measures Visit Sheet.
- 5. Gently press the PUSH end of the pulse-ox again to open the clip and release the finger.
- 6. The pulse-ox will turn off on its own.
- 7. Use an alcohol swab to gently clean the inside of the clip.
- 8. You can store it back in its blue carrying case.
- 9. If the low battery icon shows up on the display, you need to switch out the batteries.
  - a. Flip the pulse-ox over and slide off the blue battery cover.
  - b. Replace the two AAA batteries.
  - c. Replace the blue cover.



#### **Referral Protocol**

The outcomes targeted in the KidsAIR study are illnesses in children so it is anticipated that significant illness might be encountered. Epidemiologic data and other studies give evidence that such cases are few but ethically plans should be in place for field workers encountering them (RESPIRE studies, RSV statistics). In keeping with the Presidential Commission for the Study of Bioethical Issues (Bioethics Commission) in its report, Anticipate and Communicate: Ethical Management of Incidental and Secondary Findings in the Clinical, Research, and Direct-to-Consumer Contexts (http://bioethics.gov/sites/default/files/FINALAnticipateCommunicate\_PCSBI\_0.pdf), the following outline describes our protocol for management of incidental illnesses in the subjects enrolled in the KidsAIR study.

- 1. The medical resources of specific areas will be determined by participating investigators prior to collection of any field data and that list of resources will be provided to each field worker in anticipation of emergent or urgent needs. That list will include local Emergency Medical Services, physicians and health care facilities. In some specific areas, families are served by health care aides or nurses and when that is the case those persons will be the first contact for non-emergent cases.
- 2. Local healthcare providers will be contacted prior to study initiation and made aware of the nature of the study and intent of the fieldworkers.
- 3. Educational sessions will be provided to each field worker outlining signs of serious illness for the age groups being studied (World Health Organization IMCI program). Signs of illness will be categorized as life threatening (emergent), urgent, or recommended for scheduled evaluation by a health care provider. Each category of illness will initiate a different level of response.
  - a. Emergency calls will be made to the closest available emergency personnel. The field workers will stay at the home until emergency personnel arrive.
  - b. Urgent calls (non-emergency but needing care in less than 24 hours) will be made to the primary health care provider identified by the parents. Should the family have no such provider, the closest emergency room and health care provider will be contacted.
  - c. For illnesses that do not require emergent or urgent care, the parents will be advised to contact their health care provider. The field data collector will volunteer to help families make contact with appropriate health care providers. A phone call to the family will be made the following day to ensure referral has been made.
- 4. The field worker will first discuss concerns for incidental findings with the parent or care provider and they will be asked if they have a health care provider. If time allows, that person or facility will be the first notified of possible need for medical care. If the child does not have a primary care provider, a list of possible medical care providers or institutions will be provided.

#### **Referral Protocol (continued)**

Emergent signs and symptoms - call for immediate assistance to 911 local EMS

Not breathing

Cyanosis (blue coloration to the skin)

Unresponsive to stimulation

Pulseless or thread, weak pulse

Seizures

Urgent care (call to local health care aid or physician)

Difficulty breathing – retractions involving use of neck muscles and lower chest

Pulse oximetry less than 90%

Respiratory Distress - wheezing, stridor, muffled voice, difficulty speaking

Coughing up blood

Listlessness

Fever > 100.4 °F (<2 month)

> 102.2 °F (2 months – 12 months)

> 102.2 °F and ill appearing (>12 months)

Active bleeding

Stiff neck and signs of mental status change or fever

Recommend follow up with primary care provider within the next day

Wheezing not responsive to home medications but little or no distress

Prolonged fever (more than 2 days)

Prolonged cough (> 3 days)

Prolonged illness and not getting better (>1 week)

# HOME CHARACTERISTICS DATA SHEET

| Technician: | Home ID: | Winte | er (1,2,3, | etc.): |
|---|---|---|---|---|
| Sampling Dates: | Date form co | ompleted: | | |
| To be completed by an ac | dult resident on | ce at the begi | nning | of each winter. |
| 1. Number of total residents in | n home: | | | |
| 2. Number of residents young | er than 18 years of | age: | | |
| 3. Number of residents young | er than 5 years of a | .ge: | | |
| 4. Type of home: House | Mobile Home | Duplex/Apt | Other: | |
| 5. Year home built: | | | | |
| 6. Square footage of home: | | | | |
| 7. Number of floors (not incl. | bsmnt): 1 | 2 3 | | |
| 8. Number of windows: | | | | |
| 9. Number of bedrooms: | | | | |
| 10. Total number of pets: | | | | |
| 11. Total number of "furry" pe | ts: | | | |
| 12. Type of primary heating (P | lease circle ONLY | one choice that | represei | nts your most common practice): |
| Wood stove Electrical | Propane Natu | ıral gas furnace | Oil | Other: |
| 13. Type of secondary heating | (Please circle <b>ONL</b> | Y one choice th | at repres | sents your most common practice): |
| Wood stove Electrical | Propane Natu | ıral gas furnace | Oil | Other: |
| 14. Existing appliance(s): Fire | eplace Wood stor | ve Furnace | Wood | stove insert |
| 15. Wood stove model (If you i | have access, inform | nation is located | on the b | pack of the stove): |
| 16. Approximately how old is | your wood stove: | | | |
| 0-5 years old 6-10 years | ars old 11-1 | 5 years old | 16 + v | ears old |

| 17. | Is your wood | l stove EPA- | certified? | Yes | No | I don' | t know |
|---|---|---|---|---|---|---|---|
| 18. | When was th | e last time y | ou had your | chimney c | leaned? | | |
| | Less than 6 n | nonths ago | 6-12 mor | nths ago | 12-18 month | ns ago | more than 18 months ago |
| 19. | | | - | | lamp spots on<br>lings or carpet | | s inside your home other than in the |
| | Yes | No | I don't kno | w | | | |
| 20. | Has there bee | en mold or n | nildew on ar | y surfaces | inside your ho | ome in t | he last 12 months? |
| | Yes | No | I don't kno | W | | | |

# **HOME ACTIVITY LOG**

| Technician: Home ID: Winter (1,2,3,etc.): Sampling Day (1 – 6): Sampling Date: | | |
|---|---|---|
| To be completed by an adult reside | nt for each d | lay of six day sampling visit. |
| Were any of the following heating a used in the home during the sampling | | r than your woodstove, |
| <ul> <li>Gas</li> <li>Electrical</li> <li>Propane</li> <li>Oil</li> <li>Other, specify:</li> </ul> | No<br>No<br>No<br>No<br>No | Yes<br>Yes<br>Yes<br>Yes |
| Other, speerly | 110 | 103 |
| 2. Did any of the following activities o sampling period? | r conditions oc | cur in the home during the |
| • Smoking by anyone in the home (cigarette, pipe, or other) | No | Yes |
| • Incense burning | No | Yes |
| Candle burning | No | Yes |
| Kerosene/oil lamp | No | Yes |
| • Open windows | No | Yes |
| • Front door propped open | No | Yes |
| Dusting/sweeping/vacuuming | No | Yes |

# WOOD STOVE USAGE LOG

Technician:

| Wi<br>Sa | ome ID:<br>inter (1,2,3,etc.):<br>impling Dates:<br>te form completed | : | | | |
|---|---|---|---|---|---|
| | be completed mpling visit. | by an adult resid | lent at t | he end of e | ach six day |
| 1. | - | ing period, how wou<br>pical winter day (circ | - | scribe the lev | el of wood burning |
| | No burning | Light burning | Avera | ge burning | Heavy burning |
| 2. | What kind of woo | od was used or was u | sed most | frequently? F | Please choose <b>ONLY</b> one |
| | Lodgepole Pine | Ponderosa I | Pine | Fir | Larch |
| | [LIST OTHER CO | OMMON TYPES] _ | | | |
| 3. | | your wood before bu | • • | Please circle ( | <b><u>ONLY</u></b> one choice that |
| | A few days | | | Between 1 v | week and 1 month |
| | Between 1 month | and 3 months | | Between 3 n | months and 6 months |
| | Between 6 month | s and 1 year | | More than 1 | year |
| 4. | On average, how | many cords of wood | do you b | urn each year | ? cords |
| 5. | | lly acquire your woo<br>nost common practice | | e circle <u>ONL</u> | $\underline{\mathbf{Y}}$ one choice that |
| | Harvest yourself | Purchase it | | Other: | |

## **IN HOME LOG**

| Technician: |
|---------------------|
| Home ID: |
| Child ID: |
| Winter: |
| Sampling dates: |
| Sampling start time |

# To be completed by an adult resident for each participating child for each 24 hour period of six day sampling visit.

For each row, please mark the day of week (M, T, W, Th, F, Sa, Su) and whether your child was or was not home. If your child was not at home, please mark the circle indicating where your child was.

| Age of partici | ipating | child: _ |
|----------------|---------|----------|
| Child is a: | girl | boy |

| | | | | | | If not home, where? | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | Day of<br>week | Time | | | At he | ome? | school | day<br>care | relative's<br>house | friend's<br>house | other |
| 1 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 1 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 1 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 1 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 1 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 1 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 1 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 1 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 1 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 1 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 1 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 1 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 1 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 1 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 1 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 1 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |

Home ID: Child ID: Winter: Sampling dates: Sampling start time:

| | | | | | | | | If not home, where? | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| D. | Day of | | m. | | A 4 1. | 0 | | day | relative's | friend's | .4 |
| Day | week | | Time | | | ome? | school | care | house | house | other |
| 2 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 2 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 2 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 2 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 2 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 2 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 2 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 2 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 2 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 2 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 2 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 2 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 2 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 2 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 2 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 2 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |
| 3 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 3 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 3 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 3 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 3 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 3 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 3 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 3 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 3 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 3 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 3 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 3 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 3 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 3 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 3 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 3 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |

Home ID: Child ID: Winter: Sampling dates: Sampling start time:

| | | | | | | | | If not home, where? | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day of | | | | | | | day | relative's | friend's | |
| Day | week | | Time | ; | At h | ome? | school | care | house | house | other |
| 4 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 4 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 4 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 4 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 4 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 4 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 4 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 4 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 4 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 4 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 4 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 4 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 4 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 4 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 4 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 4 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |
| 5 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 5 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 5 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 5 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 5 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 5 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 5 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 5 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 5 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 5 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 5 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 5 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 5 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 5 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 5 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 5 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |

Home ID: Child ID: Winter: Sampling dates: Sampling start time:

| | | | | | | | | If not home, where? | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day of | | | | | | | day | relative's | friend's | |
| Day | week | | Time | | | ome? | school | care | house | house | other |
| 6 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 6 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 6 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 6 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 6 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 6 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 6 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 6 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 6 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 6 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 6 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 6 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 6 | | 7:00 PM | to | 8:00 PM | Y | N | | | | | |
| 6 | | 8:00 PM | to | 9:00 PM | Y | N | | | | | |
| 6 | | 9:00 PM | to | 10:00 PM | Y | N | | | | | |
| 6 | | 10:00 PM | to | 7:00 AM | Y | N | | | | | |
| 7 | | 7:00 AM | to | 8:00 AM | Y | N | | | | | |
| 7 | | 8:00 AM | to | 9:00 AM | Y | N | | | | | |
| 7 | | 9:00 AM | to | 10:00 AM | Y | N | | | | | |
| 7 | | 10:00 AM | to | 11:00 AM | Y | N | | | | | |
| 7 | | 11:00 AM | to | 12:00 PM | Y | N | | | | | |
| 7 | | 12:00 PM | to | 1:00 PM | Y | N | | | | | |
| 7 | | 1:00 PM | to | 2:00 PM | Y | N | | | | | |
| 7 | | 2:00 PM | to | 3:00 PM | Y | N | | | | | |
| 7 | | 3:00 PM | to | 4:00 PM | Y | N | | | | | |
| 7 | | 4:00 PM | to | 5:00 PM | Y | N | | | | | |
| 7 | | 5:00 PM | to | 6:00 PM | Y | N | | | | | |
| 7 | | 6:00 PM | to | 7:00 PM | Y | N | | | | | |
| 7 | _ | 7:00 PM | to | 8:00 PM | Y | N | | | | | |

## **End of Winter Questionnaires**

## **Education Homes:**

- 1. Post winter Questionnaire Education Homes
- 2. KAB Education Homes Post Winter 1 & 2 Assessment

#### **Filter Homes:**

- 1. Post winter Questionnaire Filter Homes
- 2. KAB Filter Homes Post Winter 2 Assessment

# **Post Winter Questionnaire - Education Homes**

| Home I | D: | | | Techn | ician: | | |
|---|---|---|---|---|---|---|---|
| Date: _ | | | | | | | |
| Filled o | ut by: | Mother | Father | Other: | | | |
| Please each ite | - | the followi | ng brief survey re | egarding your expo | eriences this v | vinter. Please circle your response b | elow |
| 1. | How ofte | en did you ι | use the moisture | meter during this | winter? | | |
| | Never | Once | Once a Month | Weekly | Daily | | |
| 2. | Did you s | split the wo<br>No | | reading from the f<br>Applicable | freshly cut por | tion of the log? | |
| 3. | How eas | y has it bee | n to use the moi | sture meter? | | | |
| | Difficult | Somewl | nat Difficult | Somewhat Easy | Easy | Not Applicable | |
| 4. Has the moisture meter been helpful to you this winter? | | | | | | | |
| | Not Help | | Not Very Helpfu<br>can you tell us v | | : Helpful | Very Helpful | |
| 5. | How ofte | en did you ເ | use the wood sto | ve thermometer o | during this win | <br>ter? | |
| | Never | Once | Once a Month | Weekly | Daily | | |
| 6. | How eas | y has it bee | n to use the woo | od stove thermom | eter? | | |
| | Difficult | Somewl | nat Difficult | Somewhat Eas | sy Easy | Not Applicable | |
| 7. | Has the | wood stove | thermometer be | een helpful to you | this winter? | | |
| | Not Helpful Not Very Helpful Somewhat Helpful Very Helpful If it was not helpful, can you tell us why? | | | | | | |
| 8. | How ofte | en did you ເ | use the firestarte | rs during this wint | er? | | |
| | Never | Once | Once a Month | Weekly | Daily | | |
| 9. | | | n to use the fires | | _ | | |
| | Difficult | Somewl | nat Difficult | Somewhat Eas | sy Easy | Not Applicable | |

| 10. | Have the firestarters been helpful to you this winter? | | | |
|---|---|---|---|---|
| | Not Helpful | Not Very Helpful | Somewhat Helpful | Very Helpful |
| | If it was not helpfu | If it was not helpful, can you tell us why? | | |
| 11 | Llaw often did you | wasall an watala the and | | |
| 11. | | | cational videos during thi | s winter? |
| | Never Once | Once each Month | Weekly | |
| 12. | How easy has it be | en to use the guidelines | s included in the educatio | nal videos? |
| | Difficult Somew | vhat Difficult Son | newhat Easy Easy | Not Applicable |
| 13. | Have the guidelines included in the educational videos been helpful to you this winter? | | | |
| | Not Helpful | Not Very Helpful | Somewhat Helpful | Very Helpful |
| | If it was not helpfu | I, can you tell us why? | | |
| 14. | • | | • | check in on your child's health and to ask a ful with troubleshooting issues regarding |
| | Not Helpful | Not Very Helpful | Somewhat Helpful | Very Helpful |
| | If these calls were | not helpful, can you tell | us why? | |
| 15. | Was there anything new/interesting/helpful that you learned this winter about burning more efficiently and/or cleaner with your wood stove? | | | |

## KAB - Education Homes - Post Winter 1 & 2 Assessment

| Home I | D: | | | Date: | | | |
|---|---|---|---|---|---|---|---|
| Filled o | out by: | Mother | Father | Other: | | _ | |
| There how us follow when s Please | are no<br>seful t<br>ing ite<br>you us<br>rank | o "right or w<br>he education<br>ems in terms<br>sed your woo<br>the items on | rong" answ<br>nal materia<br>of how imp<br>od stove the<br>na scale of 1 | ers to these it<br>ls and videos<br>oortant, helpfo<br>past winter.<br>l-4 | about your woodst<br>ems. This informa<br>were for you this v<br>ul, and useful the fo | tion will he<br>winter. Plea<br>ollowing su | ase rank the<br>ggestions were |
| During | g the pa | ast year how | important h | as it been: | | | |
| • | To spli | it your firewo | od in smaller | sizes (6 inches | or less in diameter)? | | _ |
| • | To stor | re your firewo | ood in a cover | red wood pile? | | | _ |
| • | To sea | son firewood | for 6-12 mor | ths before burn | ing? | | _ |
| • | To use | a moisture m | eter to test ye | our wood? | | | _ |
| • | To onl | y burn dry, se | asoned wood | l (moisture cont | ent <20%)? | | _ |
| • | To ma | intain a bed o | f ash just bel | ow the vent hole | es of the wood stove | ? | _ |
| • | To cra | ck a window/o | door on the s | ame level when | starting a fire? | | _ |
| • | To use | dry kindling, | air moveme | nt, and fire start | ers to help you | | |
| | start a | hot fire? | | | | | _ |
| • | To allo | ow small hot f | ires that burn | for 20 to 30 m | inutes to reach | | |
| | optima | al burn temper | ratures? | | | | |
| • | To use | a wood stove | thermomete | r to help you bu | ırn at | | |
| | specifi | c desired tem | peratures | | | | |
| • | To che | eck your wood | l stack 20-30 | minutes after s | tarting to burn? | | |
| • | To allo | ow the fire to l | burn for 20-3 | 0 minutes before | re refueling? | | |
| • | To not | burn items ot | ther than woo | od (e.g., trash, c | ardboard, etc.)? | | |
| • | To clea | an your flue a | nd chimney? | | | | |
| • | To con | ndition or dry | wood inside | for 2 days befor | re burning? | | |
| • | To det | ermine wood | stove model | and locate man | ual | | |

# **Post Winter Questionnaire - Filter Homes**

| Но | me ID: | | _ | Technician: | | |
|---|---|---|---|---|---|---|
| | | Mother | | Other: | | |
| | ease comple<br>low each ite | | ing brief survey r | egarding your experience | es this winter. Please | e circle your response |
| 1. | Did you us | se your Filter | unit this winter? | Yes No | | |
| 2. | Did you us | se your Filter | unit continuously | y throughout the winter? | Yes No | |
| 3. | - | not use your<br>turned on?_ | | uously, approximately ho | w many hours per w | eek did you have your |
| 4. | | etting(s) did<br>ach setting be | - | er unit when you had it tu | ırned on? Please indi | cate the percentage of |
| | High | Med | diumLow_ | | | |
| 5. | If you deci | ided not to us | se the Filter unit, v | what were the reasons? | | |
| | Noise | Cost | Appearance | Space Concerns | Inconvenience | N/A |
| | Other | | | | | |
| | Other_ | | | | | |
| 6. | Of the reas | sons above, v | which was the mos | st important reason? | | |
| | | | | | N/A | |
| 7. | Overall, do | o you think th | ne Filter unit has l | peen helpful to you and/o | or your family this wi | nter? |
| | Not Helpfu | al No | ot Very Helpful | Somewhat Helpful | Very Helpful | |

## **KAB - Filter Homes - Post Winter 2 Assessment**

| Home ID: | | | Date: | | | |
|---|---|---|---|---|---|---|
| Filled out by: | Mother | Father | Other: | | | |
| There are nyour woods are when yo Please rank | no "right or wr<br>stove usage. Pl<br>ou have used y<br>k the items on | ong" answe<br>ease rank th<br>our wood s<br>a scale of 1- | rs to these itence following it tove the past to the past to the past to the | out your woodstovens. This information of how wo years. somewhat impor | on just helps us<br>ow important tl | s understand<br>hese factors |
| During the | past two years | s how impor | tant has it bee | en: | | |
| • To sp | olit your firewoo | d in smaller s | izes (6 inches or | r less in diameter)? | | |
| • To ste | ore your firewoo | od in a covere | d wood pile? | | | |
| • To se | eason firewood f | or 6-12 month | ns before burnin | g? | | |
| • To us | se a moisture me | eter to test you | ır wood? | | | |
| • To or | nly burn dry, sea | soned wood ( | moisture conter | nt <20%)? | | |
| • To m | aintain a bed of | ash just below | v the vent holes | of the wood stove? | | |
| • To cr | ack a window/d | oor on the sar | ne level when st | tarting a fire? | | |
| | se dry kindling, a<br>a hot fire? | air movement | , and fire starter | s to help you | | |
| | low small hot final burn tempera | | For 20 to 30 min | utes to reach | | |
| • To us | se a wood stove | thermometer | to help you burr | n at | | |
| speci | fic temperatures | ? | | | | |
| • To ch | neck your wood | stack 20-30 m | ninutes after star | ting to burn? | | |
| • To al | low the fire to b | urn for 20-30 | minutes before | refueling? | | |
| • To no | ot burn items oth | er than wood | (e.g., trash, care | dboard, etc.)? | | |
| • To cl | ean your flue an | d chimney? | | | | |
| • To co | ondition or dry w | wood inside fo | or 2 days before | burning? | | |
| • To de | etermine wood s | tove model ar | nd locate manua | 1? | | |

#### **Statistical Analysis Plan**

Analysis was conducted using R version 3.6.2 (The R Foundation for Statistical Computing, Austria). We calculated descriptive statistics for continuous variables (n, mean, standard deviation [sd], minimum [min], median, maximum [max]) and categorical variables (n, percentage of total) across all study households and separately for each treatment arm and study area. We averaged indoor concentrations of PM2.5 over the 6-day sampling period for each home and for the times during which each child was reported as being at the household.

Primary analyses were conducted within three model frameworks using the Ime4 package (Bates et al. 2015): 1) intent-to-treat (ITT) framework with LRTI outcome (ITT-LRTI), 2) ITT framework with PM2.5 outcome (ITT-PM2.5), and 3) exposure-response (ER) framework with LRTI as the outcome and PM2.5 as the exposure of interest. Although LRTI cases were collected as count data, very few children had more than one LRTI, resulting in under-dispersed data that violated the assumptions of attempted Poisson and negative binomial regression models. Thus, the ITT-LRTI framework utilized mixed effects logistic regression models (using the glmer function) with presence of LRTI (yes or no) as the outcome and assigned treatment as the exposure of interest. The ITT-LRTI models included a covariate for person-time at risk to account for the wide variability of child-weeks at risk across study participants. The models also included a covariate for child age (<1 year vs. 1 to 4 years) since randomization occurred within strata of this term. A nested random term (i.e., household:cohort:area) was included in the model to account for repeated measures clustered within household, cohort, and study area. The ITT-PM2.5 framework used mixed effects linear models (using the Imer function) with mean 6-day indoor PM2.5 concentration as the outcome and assigned treatment as the exposure of interest. Models were adjusted for child age and included a nested random term of cohort:area (there were no repeated measures within household for PM2.5). Both ITT models utilized the study's randomization and were not adjusted for potential confounding variables in the primary analyses.

The ER framework utilized mixed effects logistic regression models (using the glmer function) with presence of LRTI (yes or no) as the outcome and mean 6-day indoor PM2.5 concentration as the exposure of interest. As with the ITT-LRTI models, ER models were adjusted for person-time at risk and included a nested random term (i.e., household:cohort:area) to account for repeated measures in the analysis. In addition, since the ER models did not utilize the study's randomization to help control for confounding, covariates were included in the model to adjust for potential confounders. Confounders were identified a priori through previous literature and by assessing independent associations with the exposure and outcomes of interest (Adaji et al. 2019; Mortimer et al. 2017; Noonan et al. 2019; Smith et al. 2011; Walker et al. 2021). We also used directed acyclic graphs (DAGs) to assess the direction and potential relationship between indoor PM2.5, LRTI, and covariates (Figure S3). Final ER models were adjusted for child age and sex, caregiver race and sex, household income, caregiver education, if a household resident smoked, and ambient temperature and PM2.5.

The primary ITT model framework was prespecified in our previously published methods paper (Noonan et al. 2019). We conducted a number of sensitivity analyses in all model frameworks that were specified a priori (during the initial model development when the analyst was masked to treatment arm assignment) and assessed the impact of including potential confounders in the models and using subsets of the data. We conducted sensitivity analyses by including potential confounders that had some imbalance across study arms (ITT frameworks) or by including additional potential confounders not included in the primary model (ER framework). Due to the different control treatment in AK (no filtration unit), we conducted the ITT-LRTI and ITT-PM2.5 analyses with AK households excluded from the dataset. For the ITT-LRTI and ER frameworks, we also conducted a sensitivity analysis with a dataset restricted to Winter 1 only, as this was the only winter of observation when indoor PM2.5 was sampled. For the ER framework we conducted an additional sensitivity analysis that used indoor PM2.5 when each child was at home as the primary exposure variable in place of indoor PM2.5 over the entire sampling period.

We also conducted some post hoc sensitivity analyses for the ITT-LRTI framework with other model variations to provide insight into our primary model selection and results. Specifically, we assessed models that 1) used

study area (AK, NN, WMT) as a fixed effect rather than a random nested term, 2) removed the covariate for person-time at risk, and 3) removed the random nested term for household.

We evaluated potential modification of the effect of the treatments by a priori selected child, caregiver, and home characteristics within each of the model frameworks by including interaction terms in the primary model. We assessed significance of the interaction terms using Type II Wald Chi-square tests. Model assumptions were evaluated in all analysis frameworks. Indoor PM2.5 concentrations were natural-log transformed in the ITT-PM2.5 framework, and estimates are presented as percent difference in geometric mean PM2.5.